CLINICAL TRIAL: NCT06716320
Title: Maternal Serum Insulin-Regulated Aminopeptidase (IRAP) Levels in Gestational Diabetic Pregnant Women
Brief Title: Decreased Insulin Regulated Aminopeptidase (IRAP) Levels in Gestational Diabetes Mellitus
Acronym: (IRAP)
Status: Completed | Type: Observational
Sponsor: OSMAN KÖSE, MD (Other)
Responsible Party: Sponsor-Investigator, OSMAN KÖSE, MD, assistant professor, Sakarya University
Organization: Sakarya University (Other)
Other Study IDs: E-16214662-050.01.04-28527-89
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Insulin-regulated aminopeptidase; gestational diabetes mellitus; glucose transporter 4; insulin resistance; glycated hemoglobin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group gestational diabetes mellitus, Group Healthy pregnant women: Group gestational diabetes mellitus (GDM): GDM was diagnosed according to the criteria of The International Association of Diabetes and Pregnancy Study Groups when one or more abnormal plasma glucose values were obtained (fasting ≥ 92 mg/dL, 1 h ≥ 180 mg/dL, 2 h ≥ 153 mg/dL). In pregnant women who could not achieve normoglycemia with diet, insulin treatment was started and fasting blood sugar and 1st and 2nd hour postprandial blood sugar threshold values were determined as 95 mg/dL, 140 mg/dL and 120 mg/dL, respectively.
  Group Healthy pregnant women: In the healthy pregnant women group, 40 pregnant women were considered normoglycemic because their 75-g OGTT tests matched the study group in terms of age, BMI, and gestational age. Pregnant women in this group who did not have any complications were included.
  All groups were followed until the end of birth.

SUMMARY:
This cohort study investigated whether IRAP levels could be a marker for predicting gestational diabetes mellitus. 80 women were included in the study, including the control group. The study duration was 12 months and the study was completed.

DETAILED DESCRIPTION:
In the cohort study, the study group (GDM group) consisted of 40 pregnant women diagnosed with GDM between 24-28 weeks of gestation with a 2-hour 75-g oral glucose tolerance test (OGTT). While 11 women in the GDM group received insulin treatment, 29 of them provided blood sugar regulation with diet. The 75-g OGTT tests of the 40 pregnant women in the control group were considered normoglycemic while matching with the study group in terms of age, BMI and gestational weeks, and no complications were observed in the pregnant women in this group. Pregnant women with preeclampsia, chronic hypertension, pre-gestational diabetes mellitus, any acute or chronic disease, premature birth, premature rupture of membranes (PPROM), fetal structural or chromosomal anomalies, multiple pregnancies and fetal growth restriction were not included in the study. The ELISA method determined Serum IRAP levels.

Serum IRAP levels of pregnant women were measured with enzyme-linked immunosorbent assay. Serum levels of IRAP marker were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies undergoing a 2-hour 75 g oral glucose tolerance test (OGTT) at 24 and 28 weeks of gestation.

Exclusion Criteria:

* Preeclampsia, chronic hypertension, pregestational diabetes mellitus, pregnant women with any acute or chronic disease, preterm labor, premature rupture of membranes (PPROM), fetal structural or chromosomal anomalies, multiple pregnancies, and fetal growth restriction

Ages: 21 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Singleton pregnancies undergoing a 2-hour 75 g oral glucose tolerance test (OGTT) at 24 and 28 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of serum IRAP levels | up to 1 year
  Comparison of serum IRAP levels measured during the assessment between pregnant women diagnosed with gestational diabetes mellitus (GDM) based on a 75-gram OGTT performed at 24-28 weeks of gestation and normoglycemic pregnant women.
Evaluation of serum in the pregnant women at 24-28 weeks in ng/ml. | up to 1 year
  For IRAP measurements, blood samples taken between weeks 24 and 28 were centrifuged and the serum was separated and stored at -80 ° C until the day of the study. On the day of the study, all samples were thawed at the same time and included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Osman köse, ass. Prof., Study Director — Sakarya University Faculty of Medicine
Locations (1):
- Sakarya University Faculty of Medicine, Adapazarı, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) will be shared. Data to be shared will include age, gender, and clinical outcomes. Data will be shared with appropriate researchers after the results of the study are published. Data requests will be evaluated within the framework of relevant ethical rules.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared with appropriate researchers after the results of the study are published.
Access Criteria: The full dataset or specific requested data will be accessible to researchers conducting academic research upon request or through data-sharing platforms for a period of 3 years

REFERENCES:
- [Result] Vear A, Thalmann C, Youngs K, Hannan N, Gaspari T, Chai SY. Development of a sandwich ELISA to detect circulating, soluble IRAP as a potential disease biomarker. Sci Rep. 2023 Nov 24;13(1):17565. doi: 10.1038/s41598-023-44038-1. PMID 38001104